CLINICAL TRIAL: NCT01982175
Title: A Multi-center, Open, Prospective, Phase II Study of Recombinant Humanized Anti-CD52 Monoclonal Antibody Injection in Patients With Relapse and Refractory B-cell Chronic Lymphocytic Leukemia
Brief Title: Phase II Clinical Trial of Alemtuzumab to Treat B-cell Chronic Lymphocytic Leukemia
Acronym: CLL004
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: recruiting difficulties
Sponsor: Shanghai Zhangjiang Biotechnology Limited Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMAB004
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
Keywords: Alemtuzumab; B-cell chronic lymphocytic leukemia; CD52
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alemtuzumab (Experimental): Patients receive Alemtuzumab escalated from initial dose of 3mg/day then 10mg/day and up to 30mg/day by intravenous infusion(if tolerated). when stable dose of 30mg/day is tolerated, Alemtuzumab is administrated at 30mg by IV infusion 3 times per week for up to 12 weeks (including escalation and stable dose period). After completion of 12 weeks treatment, or discontinuation of treatment within 12 weeks due to disease progression, patients will be visited every 3 months up to 1 year from enrollment or to death, whichever occurs first.
  Interventions: Biological: Alemtuzumab

INTERVENTIONS:
Biological: Alemtuzumab — Escalation Phase: Initial Doses of Alemtuzumab 3mg/day by intravenous(IV) infusion until tolerated, then Alemtuzumab 10mg/day IV infusion until tolerated, then Alemtuzumab 30mg IV infusion until tolerated.
  Escalation to 30mg/day should be accomplished in 3~7 days.
  Stable dose Phase: Once 30mg/day infusion of Alemtuzumab was tolerated, then continue 3 times per week. The total duration of Alemtuzumab therapy including escalation and stable dose phase is 12 weeks.
  More than 30mg daily or 90mg weekly dose is prohibited
  --------------------------------------------------------------------------------
  Other Names: Recombinant Humanized Anti-CD52 Mab

SUMMARY:
This is a phase II, prospective, multicenter, open-label study to evaluate the efficacy and safety of Alemtuzumab in patients with relapse and refractory B-cell chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* An established diagnosis of B-cell chronic lymphocytic leukemia(B-CLL)
* Meet criteria of relapsed or refractory CLL
* Presence of one or more measurable lesions
* ECOG Score 0-1
* Life expectancy > 3 months
* Female patients with childbearing potential must have a negative serum pregnancy test, male and female patients must agree to use an effective contraceptive method while on study treatment, and for a minimum 1 year following study therapy.

Exclusion Criteria:

* Less than 2 weeks from prior anti-cancer therapy.
* Allergic to the antibody or any component of the investigational product.
* Other severe, concurrent diseases, including mental disorders, serious cardiac functional capacity (Class III or IV), uncontrolled diabetes.
* Use of investigational agents rather than Alemtuzumab.
* Active systematic infection or major organ malfunction requiring treatment.
* Serum total bilirubin greater than or equal to 1.5 times upper limits of normal; or Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) greater than or equal to 2.5 times upper limits of normal ( no liver metastases); or ALT and/or AST greater than or equal to 5 times upper limits of normal (liver metastases).
* Blood urea nitrogen(BUN) greater than or equal to 1.5 times upper limits of normal or Serum creatinine greater than or equal to 1.5 times upper limits of normal.
* White blood cell(WBC) count< 3.5×109/L or Absolute neutrophil count(ANC)<1.5×109/L or platelet count<75×109/L or Hemoglobin<80g/L.
* Human immunodeficiency virus (HIV) positive.
* Active hepatitis or a history of prior viral hepatitis B or C, or positive hepatitis B serologies without prior immunization.
* Pregnant or nursing women.
* Known central nervous system(CNS) metastases with B-CLL.
* Active secondary malignancy.
* cytomegalovirus(CMV) positive or immunodeficiency disease or after stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-07; Primary Completion 2021-02 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 1 year
  Objective Response Rate was defined as the proportion of patients who have CR, PR during the study as evaluated according to National Comprehensive Cancer Network(NCCN) guideline 2010 response criteria. Response categories include Complete Response(CR) and Partial Response(PR).
  ORR=CR+PR

SECONDARY OUTCOMES:
Progression-Free Survival | up to 1 year
  Progression-Free Survival was defined as the time from randomization to disease progression (PD) or death due to any cause, whichever comes first.
Disease Control Rate(DCR) | up to 1 year
  Patients were evaluated according to National Comprehensive Cancer Network(NCCN) guideline 2010 response criteria. The best response observed during the study is summarized. Response categories include Complete Response(CR), Partial Response(PR) and Stable Disease(SD).
  DCR=CR+PR+SD
Duration of Response(DOR) | up to 1 year
  Duration of response was analyzed for patients who achieved a complete release(CR) or partial release(PR) and was defined as the time from the first date of documented response to the date of disease progression or death due to any cause.
Overall Survival | up to 1 year
  Overall Survival was defined as the duration from randomization to death due to any cause.
Summary of patients with Adverse Events(AEs) | up to 1 year
  Analysis of patients with adverse experiences according to CTCAE Version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, M.D., Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China